CLINICAL TRIAL: NCT00408863
Title: A Multinational, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Trial to Investigate Safety and Efficacy of Tibolone (Org OD14) in Women With Climacteric Symptoms and a History of Breast Cancer
Brief Title: Livial Intervention Following Breast Cancer; Efficacy, Recurrence and Tolerability Endpoints (LIBERATE)(COMPLETED)(P05885)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P05885; 32974
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer; Climacteric Symptoms
Keywords: Breast cancer; Tibolone; Climacteric symptoms
MeSH Terms: conditions — Breast Neoplasms | interventions — tibolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tibolone (Active Comparator): Tibolone 2.5 mg/day
  Interventions: Drug: tibolone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tibolone — tibolone 2.5 mg/day
  Other Names: OD-14
  Arms: Tibolone
Drug: placebo
  Arms: Placebo

SUMMARY:
Postmenopausal women with a history of breast cancer often suffer from climacteric symptoms such as hot flushes and sweating episodes. Conventional hormone therapy is not allowed in such patients because there are indications that hormones may cause breast cancer to recur.

Tibolone is a steroid with estrogenic, progestogenic and androgenic activity and is registered for treatment of climacteric complaints. Tibolone has a pharmacologic and clinical profile that is different from conventional hormones. In contrast to conventional hormones, tibolone does not increase breast density and causes less breast pain.

The LIBERATE study is a study in which the safety and efficacy of tibolone has been investigated in postmenopausal women that have been treated for breast cancer.

DETAILED DESCRIPTION:
A growing proportion of women diagnosed with early stage breast cancer seek help with vasomotor and sexual complaints. Frequently, these symptoms result from adjuvant cancer treatment, irrespectively whether this is hormonal (e.g. tamoxifen, aromatase inhibitors), cytotoxic, or surgical (oophorectomy) in nature. Estrogen-containing hormone therapy is effective, but considered unsafe. Non-hormonal therapy is less effective. Tibolone, which does not increase mammographic breast density, has proven to be effective and thus could be an important treatment option for women persistently seeking help.

The objective of this trial is to demonstrate safety, efficacy and tolerability of oral 2.5 mg tibolone daily in breast cancer patients, who, after surgery, have no evidence of disease and who suffer from climacteric complaints. Primary study endpoint is breast cancer recurrence, including primary contralateral breast cancer. Secondary outcome variables include menopausal symptoms, bone mineral density and health-related quality of life.

Patients were eligible for this study when they had been surgically treated within the previous 5 years for histologically confirmed T1-3, N0-2, M0 breast cancer and had to have vasomotor symptoms, with a last menstruation at least 12 months before (or bilateral oophorectomy).

The LIBERATE Trial has been designed to show non-inferiority of tibolone compared to placebo. Adequate sample size was estimated to be at least 1500 subjects in each arm, assuming a breast cancer recurrence rate of 5% per year in the first 3 years and an dropout rate of 5% per year.

The LIBERATE Study has successfully included the appropriate number of women with the proper risk profile so that significant results can be obtained in relation to safety and efficacy of tibolone in breast cancer patients with menopausal complaints.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed and surgically treated invasive breast carcinoma (T1/2/3 N0/1/2 M0), irrespective of hormonal (estrogen/progestogen) receptor status.
* Last menstrual bleeding at least 12 months before the start of the study or ovariectomized or hysterectomized or currently being treated with gonadotropin releasing hormone analogs.
* Vasomotor symptoms whether related to natural menopause, ovariectomy, or to breast cancer therapy (chemotherapy, tamoxifen, aromatase inhibitors or other anticancer therapy).
* In subjects with an intact uterus, a 'normal' endometrium, defined as:

  1. in tamoxifen users: absence of endometrial polyps
  2. in non-tamoxifen users: double layer endometrial thickness <=4 mm as assessed by TVUS or double layer endometrial thickness >4 mm and <=8 mm as assessed by TVUS plus an endometrial biopsy result of inactive/atrophic.
* Voluntary written informed consent and willing and able to make reasonable efforts to meet all clinical trial requirements.

Exclusion Criteria:

* Age >75 years at baseline.
* Ductal carcinoma in situ (DCIS) of the breast without the existence of invasive breast carcinoma.
* Invasive breast carcinoma having a tumor of any size with direct extension to chest wall or skin (T4) and/or having metastasis to ipsilateral mammary lymph node(s) (N3) and/or having presence of distant metastasis (M1).
* Surgical treatment of the primary breast cancer >5 years ago.
* History or presence of residual or recurrent breast cancer.
* History or presence of endometrial cancer.
* History or presence of any other malignancy (besides breast cancer and endometrial cancer) within the past 5 years, except for adequately treated basal cell carcinoma of the skin.
* Diagnostic findings suspicious for any malignancy.
* Double layer endometrial thickness >8 mm as assessed by TVUS in subjects not being treated with tamoxifen.
* Final diagnosis of endometrial biopsy different from inactive/atrophic
* Existence of endometrial polyps as demonstrated by TVUS.
* Undiagnosed vaginal bleeding.
* Abnormal cervical smear (corresponding to PAP IIb or higher)
* Any previous or current unopposed estrogen administration in women with an intact uterus (occasional use of estrogen-containing vaginal cream was allowed after an appropriate washout period - see below).
* Use of systemic estrogens and/or progestogens (including intra-uterine progestogen therapy) and/or tibolone and/or phytoestrogens within 8 weeks prior to baseline; use of transdermal hormone therapy and/or local estrogen applications and/or non-hormonal medication for vasomotor symptoms within 4 weeks prior to baseline.
* Use of progestogen implants or injections and/or estrogen/progestogen injectable therapy within the past 6 months.
* Use of estrogen implants or injections within the past 5 years.
* Use of raloxifene hydrochloride and/or any non-registered investigational drug within the last 8 weeks.
* Active deep vein thrombosis, thromboembolic disorders, or a documented history of these conditions.
* Severe liver disorders.
* Abnormal laboratory values considered to be clinically relevant by the investigator.
* Any disease or condition that is clinically relevant and which, in the opinion of the investigator, would jeopardize the subject's well-being during the course of the trial.
* Known hypersensitivity to tibolone or any of its components
* Known or suspected pregnancy
* Age <40 years at baseline and planned breast cancer therapy <2 years after baseline

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3148 (Actual)
Dates: Start 2002-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To show non-inferiority in breast cancer recurrence of tibolone 2.5 mg versus placebo in women with climacteric symptoms who have been surgically treated for primary breast cancer within the last 5 years | At clinical completion

SECONDARY OUTCOMES:
Secondary outcome variables include overall survival, menopausal symptoms, bone mineral density and health-related quality of life. | At clinical completion

REFERENCES:
- [Background] Kenemans P, Kubista E, Foidart JM, Yip CH, von Schoultz B, Sismondi P, Vassilopoulou-Sellin R, Beckmann MW, Bundred NJ, Egberts J, van Os S, Planellas J. Safety of tibolone in the treatment of vasomotor symptoms in breast cancer patients--design and baseline data 'LIBERATE' trial. Breast. 2007 Dec;16 Suppl 2:S182-9. doi: 10.1016/j.breast.2007.07.028. PMID 17983942
- [Derived] Lara LA, Cartagena-Ramos D, Figueiredo JB, Rosa-E-Silva ACJ, Ferriani RA, Martins WP, Fuentealba-Torres M. Hormone therapy for sexual function in perimenopausal and postmenopausal women. Cochrane Database Syst Rev. 2023 Aug 24;8(8):CD009672. doi: 10.1002/14651858.CD009672.pub3. PMID 37619252
- [Derived] Sismondi P, Kimmig R, Kubista E, Biglia N, Egberts J, Mulder R, Planellas J, Moggio G, Mol-Arts M, Kenemans P. Effects of tibolone on climacteric symptoms and quality of life in breast cancer patients--data from LIBERATE trial. Maturitas. 2011 Dec;70(4):365-72. doi: 10.1016/j.maturitas.2011.09.003. Epub 2011 Oct 26. PMID 22030384
- [Derived] Kenemans P, Bundred NJ, Foidart JM, Kubista E, von Schoultz B, Sismondi P, Vassilopoulou-Sellin R, Yip CH, Egberts J, Mol-Arts M, Mulder R, van Os S, Beckmann MW; LIBERATE Study Group. Safety and efficacy of tibolone in breast-cancer patients with vasomotor symptoms: a double-blind, randomised, non-inferiority trial. Lancet Oncol. 2009 Feb;10(2):135-46. doi: 10.1016/S1470-2045(08)70341-3. Epub 2009 Jan 23. PMID 19167925